CLINICAL TRIAL: NCT00102947
Title: An Open Label Phase 4 Trial to Further Evaluate the Pharmacokinetic Profile of Intravenous Daptomycin, and a Comparison of the Safety and Efficacy of Daptomycin Versus Comparator in the Treatment of Adult Patients With Renal Impairment and Complicated Skin and Skin Structure Infections Due, at Least in Part, to Gram-positive Bacteria
Brief Title: Daptomycin in the Treatment of Patients With Renal Insufficiency and Complicated Skin and Skin Structure Infections
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3009-020; DAP-REN-03-06 (Other: Cubist Study Number)
Record Dates: First submitted 2005-02-04; First posted 2005-02-07 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Soft Tissue Infections
Keywords: renal impairment; daptomycin; Cubist; complicated skin and skin structure infections
MeSH Terms: conditions — Soft Tissue Infections; Renal Insufficiency | interventions — Daptomycin

INTERVENTIONS:
Drug: daptomycin (up to 14 days)

SUMMARY:
This is a Phase 4, randomized, open-label, multicenter, comparative study designed to further evaluate the pharmacokinetics of intravenous (i.v.) daptomycin and the safety and efficacy of daptomycin relative to comparator in the treatment of complicated skin and skin structure infections in patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria: - Moderate to end-stage renal impairment - A diagnosis of complicated skin and skin structure infection known or suspected to be due to susceptible Gram-positive bacteria based on positive Gram stain - A diagnosis of bacterial skin and skin structure infection in the presence of some complicating factor Exclusion Criteria: - Known bacteremia, osteomyelitis or endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To obtain additional pharmacokinetic data (on dosing days) on intravenous daptomycin in patients with complicated skin and skin structure infections and renal impairment

SECONDARY OUTCOMES:
To compare the safety and efficacy of daptomycin to comparator in patients with complicated skin and skin structure infections and renal impairment at 14 to 21 days after last dose

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Harbor UCLA Medical Center, Torrance, California
  - Tampa General Hospital, Tampa, Florida
  - Joseph M. Still Research Institute, Augusta, Georgia
  - Infectious Diseases Minneapolis-LTD, Minneapolis, Minnesota
  - Upstate Clinical Research Associates, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - AllTrials Clinical Research, Winston-Salem, North Carolina
  - Riverside Methodist Hospital, Columbus, Ohio
  - Wright State University/Veterans Affairs Medical Center, Dayton, Ohio
  - ID Clinical Research, Toledo, Ohio
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - The Reading Hospital and Medical Center, West Reading, Pennsylvania